CLINICAL TRIAL: NCT04950335
Title: Comparison of Autologous Osteoperiosteal and Osteochondral Transplantation for the Treatment of Medial Large Cystic Osteochondral Lesions of the Talus
Brief Title: Comparison of AOCT and AOPT for the Treatment of Medial Large Cystic OLT
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021055
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Osteochondral Lesions of the Talus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AOPT: patients underwent AOPT to treat large cystic OLTs (>10mm)
  Interventions: Procedure: AOPT
- AOCT: patients underwent AOCT to treat large cystic OLTs (>10mm)
  Interventions: Procedure: AOCT

INTERVENTIONS:
Procedure: AOPT — The Osteochondral Autograft Transplant System (Arthrex) was used to create donor plugs. Osteoperiosteal grafts were harvested from the ipsilateral anterior superior iliac spine.
  Groups: AOPT
Procedure: AOCT — Osteochondral grafts were harvested from the non-weight-bearing zone of the ipsilateral anterolateral distal femur.
  Groups: AOCT

SUMMARY:
Autologous osteoperiosteal transplantation using tissue harvested from the iliac crest is used to treat large cystic osteochondral lesions of the talus. This study is to compare clinical and radiological outcomes between patients undergoing AOPT and those undergoing AOCT for large cystic OLTs.

DETAILED DESCRIPTION:
From March 2015 to March 2018, 23 patients who underwent AOPT and 23 patients who underwent AOCT to treat large cystic OLTs (>10mm) were retrospectively evaluated. For comparability, the two groups were matched based on their demographics, including sex, age, body mass index, side of injury, follow-up period, and the preoperative cyst volume. Clinical outcomes were assessed using the visual analog scale (VAS), the American Orthopaedic Foot & Ankle Society (AOFAS) score, and the Tegner score. Donor-site morbidity was recorded according to the symptoms, including pain, stiffness, swelling and discomfort. Radiological outcomes were evaluated using the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART) score, and the International Cartilage Repair Society (ICRS) score was obtained during second-look surgery.

ELIGIBILITY:
Inclusion Criteria:

* presence of medial large cystic OLTs (>10 mm in diameter) confirmed by preoperative magnetic resonance imaging (MRI)
* patients who underwent either primary AOPT or AOCT

Exclusion Criteria:

* small cystic OLTs
* ankle osteoarthritis
* ankle pigmented villonodular synovitis
* prior surgery on the ipsilateral ankle
* injuries or relevant trauma to the affected ankle after surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptomatic OLTs who underwent AOPT or AOCTvat our sports medicine institute between March, 2015 and March, 2018
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
MOCART | two years after sugery
  the Magnetic Resonance Observation of Cartilage Repair Tissue score

SECONDARY OUTCOMES:
VAS | pre-surgery, two years after sugery
  the visual analog scale
Tegner | pre-surgery, two years after sugery
  the Tegner score
AOFAS | pre-surgery, two years after sugery
  American Orthopaedic Foot & Ankle Society score
ICRS | one year after sugery
  the International Cartilage Repair Society score

CONTACTS AND LOCATIONS:
Overall Officials: Qinwei Guo, MD, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No